CLINICAL TRIAL: NCT01396330
Title: Effect of Prolonged Mental Stress During Safe Driving Training Courses on Glucose Control in Patients With Diabetes Mellitus Type 2
Brief Title: Effect of Mental Stress on Glucose Control in Patients With Diabetes Mellitus
Acronym: EMSOD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: Kantonsspital Frauenfeld (Other)
Responsible Party: Principal Investigator, Heiko Uthoff, MD, University Hospital, Basel, Switzerland
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: EMSOD
Record Dates: First submitted 2011-07-12; First posted 2011-07-18 (Estimated); Last update posted 2012-02-29 (Estimated); Status verified 2012-02

CONDITIONS: Diabetes Mellitus; Mental Stress
MeSH Terms: conditions — Diabetes Mellitus; Stress, Psychological

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Stress (Other)
  Interventions: Behavioral: stress

INTERVENTIONS:
Behavioral: stress — 3 professional safe drive training courses each lasting 30 minutes

SUMMARY:
Introduction Stress is part of the investigators daily life, and means to cope with it allow adaptation and survival. To this end, physiological pathways are activated, including neuroendocrine, cardiovascular and metabolic responses. In short term, the majority of consequences are beneficial, in the long run, however, chronic psychosocial stress may constitute an increased risk for coronary heart disease, type 2 diabetes, and disability.

Acute mental stress induces an exaggerated release of stress hormones e.g. catecholamine and cortisol which are thought not only to increase heart rate (HR) and blood pressure (BP) but also to increase blood glucose levels. In clinical practice, patients and health care providers are often confronted with questions concerning psychological stress as a possible reason for glucose fluctuations. Whether stress itself or poor treatment adherence is responsible for the altered glucose control remains often controversial. Differences in the inter- and intraindividual response to stress have been suggested, but only a few small studies have addressed the effect of acute psychological stress on glucose control in patients with diabetes. Patients with type 2 diabetes may overestimate the effect of acute psychological stress on glucose control but further studies are clearly needed to definitely exclude or confirm a relevant effect of stress on the glucose control in diabetic patients. For example, effects of longer lasting or repetitive events of psychological stress on glucose concentrations still remain elusive. The aim of the present study was therefore to investigate the effect of prolonged psychological stress by means of repetitive safe driving training courses on glucose control in patients with diabetes.

Patients and Methods Forty patients with type 1 or insulin-treated type 2 diabetes attending the outpatient-clinic of the Kantonsspital Frauenfeld or University Hospital of Zurich for regular visits are invited to participate. Included are patients on any oral glucose-lowering treatment and at least one daily injection of insulin, a valid driver license and written informed consent given. Exclusion criteria are diabetes duration <2 years, pregnancy, unstable coronary artery disease, limited visual acuity or unstable proliferative diabetic retinopathy, uncontrolled hypertension (BP >160/95mmHg) and pituitary or adrenal disease. The Ethics committee of the Kanton Thurgau approved the protocol and the study conform to the principles outlined in the Declaration of Helsinki.

Study protocol Each patient completes a control and a stress testing day which takes place consecutively in a randomized order. Randomization is performed by an uninvolved third person. The study is carried out at the driving training area of the Touring Club Switzerland at Hinwil. Patients are advised to have lunch before 12:00 a.m. and to abstain from food thenceforth. Drinking mineral water remains allowed during the entire study days, and the patients have to take their basal insulin and other medication as usual. Patients are advised to arrive at the driving training area between 2:30 and 3:00 p.m. At arrival, a capillary glucose measurement is carried out, and glucose concentrations ≥10mmol/l are corrected with short-acting insulin analogues (glucose target 6 - 8mmol/l). Subsequently, no additional adjustment with insulin is allowed during the study. Glucose concentrations ≤4mmol/l are always corrected with administration of 10g carbohydrate (DextroEnergy® or orange juice). On both study days, patients ingest a standard meal at 4:45 p.m. (i.e. 15min before the driving training). Immediately after the meal, short-acting insulin is injected in knowledge of the carbohydrate content (same dose on both days) or oral antidiabetics are ingested as usual. Measurements of capillary and plasma glucose concentration, blood pressure, heart rate, stress perception and salivary cortisol concentration are carried out in regular intervals between 4 and 9 p.m. on both study days.

On the control day, patients are placed in a quiet room and are permitted to read. They also have the possibility to leave the room and stay on a balcony.

On the stress testing day, patients complete a driving training with their car between 5 and 7 p.m. The driving training consists of 3 consecutive exercises: first, a slalom track on dry and wet asphalt, secondly, a full braking exercise with water obstacles. Thirdly, the car is hurled around by a mechanical plate and the patients has to regain control over it.

ELIGIBILITY:
Inclusion Criteria:

* diabetes mellitus type 1 and type 2
* stable glucose control
* valid driver license
* written informed consent

Exclusion Criteria:

* pregnancy
* unstable coronary artery disease
* limited visual acuity or unstable proliferative diabetic retinopathy
* uncontrolled hypertension (BP >160/95mmHg).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2011-09; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Mean and maximum change from baseline in glucose level (mmol/l) | within 240 minutes after stress
  Glucose level will be measured before and every 15-30 minutes after stress application for up to 240 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Peter Wiesli, MD, Principal Investigator — Kantonsspital Frauenfeld; Heiko Uthoff, MD, Principal Investigator — University Hospital, Basel, Switzerland
Locations (1):
- Kantonsspital Frauenfeld, Frauenfeld, Switzerland